CLINICAL TRIAL: NCT02499822
Title: Short - Medium and Long Term Blood Pressure Variability in Essential Hypertensive Patients Treated With Nifedipine GITS or Ramipril - a Randomized Trial
Brief Title: REducing Blood Pressure Variability in Essential Hypertension With RAmipril vErsus Nifedipine GITS Trial
Acronym: REVERENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09F401
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Hypertension; High Blood Pressure Variability
Keywords: Hypertension; Blood pressure variability; Home systolic blood pressure; Organ damage; Nifedipine GITS; Ramipril
MeSH Terms: conditions — Hypertension | interventions — Ramipril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine GITS 30 mg slow release (Experimental): Nifedipine GITS 30 mg slow release in tablets.
  Interventions: Drug: Nifedipine GITS
- Ramipril 10 mg (Experimental): Ramipril 10 mg in tablets.
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Nifedipine GITS — Commercially available drug formulations are used. Study medication will be assumed in a single morning (7-10 a.m.) administration per os.
  Arms: Nifedipine GITS 30 mg slow release
Drug: Ramipril — Commercially available drug formulations are used. Study medication will be assumed in a single morning (7-10 a.m.) administration per os.
  Arms: Ramipril 10 mg

SUMMARY:
The purpose of this study is

1. to compare the effects of nifedipine GITS and ramipril on blood pressure variability in subjects with elevated blood pressure variability.
2. to assess whether the degree of treatment-induced changes in blood pressure variability, is related to the degree of regression (or progression) of organ damage in heart, kidneys and carotid arteries.

DETAILED DESCRIPTION:
Elevated blood pressure variability (BPV) is associated with adverse cardiovascular outcomes and organ damage in hypertensive subjects. An antihypertensive treatment able to reduce BPV independently of BP lowering effect might thus provide additional protection in terms of cardiovascular risk in subjects with elevated BPV, independently on its effect of BP itself. However, data on the effects of different classes of antihypertensive drugs on BPV are limited and inconsistent. Some studies have suggested a possible usefulness of calcium antagonists in this setting. Based on the above considerations the investigators hypothesize that a calcium channel blocker nifedipine GITS, will provide a greater BPV lowering effect, when compared with ramipril, independently from the reduction in mean BP level. Based on the above considerations, the primary objective of this study is to compare the effects of nifedipine GITS and ramipril on different estimates of BPV (24 h BPV, home BPV, and visit-to-visit BPV) in subjects with elevated BPV. The secondary objective is to assess whether the degree of treatment-induced changes in BPV, is related to the degree of regression (or progression) of organ damage, after accounting for mean BP reduction by treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects
* Age 35-75 years
* Clinic systolic BP ≥140 mmHg and/or diastolic BP ≥ 90 mmHg (under no antihypertensive treatment)
* Daytime BP on ambulatory BP monitoring (ABPM) ≥135 mmHg systolic and/or ≥85 mmHg diastolic (under no antihypertensive treatment)
* Home SBP standard deviation (SD) >7 mmHg and/or daytime ambulatory SBP SD >12 mmHg
* Patients may be included if untreated or, if treated with one antihypertensive drug or two drugs in low doses, after 2 weeks' washout period
* Written informed consent to participate in the study

Exclusion Criteria:

* Subjects treated with ≥ 2 antihypertensive drugs (except those on two drugs in low doses)
* Treated subjects with on-treatment clinic BP ≥160 mmHg systolic and/or 100 mmHg diastolic
* Treated antihypertensive subjects in whom withdrawal of treatment is deemed unethical by the investigator (e.g. because of the existence of compelling indications other than hypertension for continuous use of previously used antihypertensive agent)
* Contraindications to study treatments as detailed in the relative Summaries of Medical Product Characteristics for ramipril (hypersensitivity to ramipril or any of the excipients or any other ACE inhibitor, history of angioneurotic oedema, extracorporeal treatments leading to contact of blood with negatively charged surfaces, significant bilateral renal artery stenosis or renal artery stenosis in a single functioning kidney, second and third trimesters of pregnancy, lactation, haemodynamically relevant renal artery stenosis, hypotensive or haemodynamically unstable patients) or nifedipine GITS (known hypersensitivity to nifedipine or to any of the excipients, pregnancy before week 20 and during breastfeeding, cardiovascular shock, concomitant treatment with rifampicin, patients with a Kock pouch)
* Cardiovascular diseases other than hypertension (coronary heart disease, heart failure or left ventricular systolic dysfunction of any degree, atrial fibrillation or frequent arrhythmias, valvular or congenital heart disease, cardiomyopathies, cerebrovascular disease, peripheral artery disease, aortic aneurysm)
* Chronic kidney disease
* Suspected or confirmed secondary hypertension
* Diabetes mellitus
* Subjects with conditions other than those mentioned above, where compelling indications for the use of any specific class of antihypertensive medication exist, according to current (e.g. European Society of Cardiology) guidelines
* Other conditions deemed relevant by the investigator (including respiratory disorders, liver disease, renal disease, thyroid disorders)
* BMI ≥35 kg/m2
* Known severe obstructive sleep apnea (apnea-hypopnea index > 30 or use of CPAP)
* Premenopausal women not using effective contraceptive methods
* Elevated probability of noncompliance with the study procedures

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-10; Primary Completion 2020-07-03 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Variability (standard deviation) of home systolic blood pressure at final visit | After 10 weeks of study treatment

SECONDARY OUTCOMES:
Variability (standard deviation) of home diastolic blood pressure measured at final visit | At baseline and after 10 weeks of study treatment
Short term 24h variability of systolic blood pressure at final visit (24h weighted standard deviation) | At baseline and after 10 weeks of study treatment
Short term 24h variability of diastolic blood pressure at final visit (24h weighted standard deviation) | At baseline and after 10 weeks of study treatment
Visit-to-visit variability (standard deviation) of systolic blood pressure assessed over the three last visits | At baseline and after 6, 8 and 10 weeks of study treatment
Visit-to-visit variability (standard deviation) of diastolic blood pressure assessed over the three last visits | At baseline and after 6, 8 and 10 weeks of study treatment
Mean 24 hour systolic blood pressure at final visit | At baseline and after 10 weeks of study treatment
Mean 24 hour diastolic blood pressure at final visit | At baseline and after 10 weeks of study treatment
Sokolow index at the end of the extension study | At baseline and after 12 months of study treatment
Cornell voltage duration index at the end of the extension study | At baseline and after 12 months of study treatment
Left ventricular mass index at the end of the extension study | At baseline and after 12 months of study treatment
Microalbuminuria (albumin-creatinine ratio) at the end of the extension study | At baseline and after 12 months of study treatment
Estimated glomerular filtration rate (eGFR, by CKD-EPI formula) at the end of the extension study | At baseline and after 12 months of study treatment
Carotid-femoral pulse wave velocity (cfPWV) at the end of the extension study | At baseline and after 12 months of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Parati, MD, Principal Investigator — Istituto Auxologico Italiano - Milan, Italy
Locations (3):
- Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital Shanghai Institute of Hypertension, Shanghai Jiaotong University School of Medicine, Shanghai, China
- Hypertension Center, Third University Department of Medicine, Sotiria Hospital, Athens, Greece
- Istituto Auxologico Italiano, Milan, Italy

REFERENCES:
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Parati G, Ochoa JE, Lombardi C, Bilo G. Assessment and management of blood-pressure variability. Nat Rev Cardiol. 2013 Mar;10(3):143-55. doi: 10.1038/nrcardio.2013.1. Epub 2013 Feb 12. PMID 23399972
- [Background] Liu JG, Xu LP, Chu ZX, Miao CY, Su DF. Contribution of blood pressure variability to the effect of nitrendipine on end-organ damage in spontaneously hypertensive rats. J Hypertens. 2003 Oct;21(10):1961-7. doi: 10.1097/00004872-200310000-00025. PMID 14508204
- [Background] Rothwell PM, Howard SC, Dolan E, O'Brien E, Dobson JE, Dahlof B, Sever PS, Poulter NR. Prognostic significance of visit-to-visit variability, maximum systolic blood pressure, and episodic hypertension. Lancet. 2010 Mar 13;375(9718):895-905. doi: 10.1016/S0140-6736(10)60308-X. PMID 20226988
- [Background] Webb AJ, Fischer U, Mehta Z, Rothwell PM. Effects of antihypertensive-drug class on interindividual variation in blood pressure and risk of stroke: a systematic review and meta-analysis. Lancet. 2010 Mar 13;375(9718):906-15. doi: 10.1016/S0140-6736(10)60235-8. PMID 20226989
- [Background] Ushigome E, Fukui M, Hamaguchi M, Tanaka T, Atsuta H, Ohnishi M, Oda Y, Yamazaki M, Hasegawa G, Nakamura N. Beneficial effect of calcium channel blockers on home blood pressure variability in the morning in patients with type 2 diabetes. J Diabetes Investig. 2013 Jul 8;4(4):399-404. doi: 10.1111/jdi.12052. Epub 2013 Mar 4. PMID 24843686
- [Background] Wang JG, Yan P, Jeffers BW. Effects of amlodipine and other classes of antihypertensive drugs on long-term blood pressure variability: evidence from randomized controlled trials. J Am Soc Hypertens. 2014 May;8(5):340-9. doi: 10.1016/j.jash.2014.02.004. Epub 2014 Feb 15. PMID 24685006
- [Background] Levi-Marpillat N, Macquin-Mavier I, Tropeano AI, Parati G, Maison P. Antihypertensive drug classes have different effects on short-term blood pressure variability in essential hypertension. Hypertens Res. 2014 Jun;37(6):585-90. doi: 10.1038/hr.2014.33. Epub 2014 Mar 27. PMID 24671016
- [Background] Mancia G, Facchetti R, Parati G, Zanchetti A. Visit-to-visit blood pressure variability in the European Lacidipine Study on Atherosclerosis: methodological aspects and effects of antihypertensive treatment. J Hypertens. 2012 Jun;30(6):1241-51. doi: 10.1097/HJH.0b013e32835339ac. PMID 22499291
- [Background] Matsui Y, O'Rourke MF, Hoshide S, Ishikawa J, Shimada K, Kario K. Combined effect of angiotensin II receptor blocker and either a calcium channel blocker or diuretic on day-by-day variability of home blood pressure: the Japan Combined Treatment With Olmesartan and a Calcium-Channel Blocker Versus Olmesartan and Diuretics Randomized Efficacy Study. Hypertension. 2012 Jun;59(6):1132-8. doi: 10.1161/HYPERTENSIONAHA.111.189217. Epub 2012 Apr 30. PMID 22547439
- [Derived] Zhang W, Liu CY, Bilo G, Soranna D, Zambon A, Kyriakoulis KG, Kollias A, Ceravolo I, Cassago S, Pengo MF, Destounis A, Stergiou GS, Wang JG, Parati G. A Randomized Controlled Trial on the Efficacy and Safety of a Calcium-Channel Blocker and an Angiotensin-Converting Enzyme Inhibitor in Chinese and European Patients with Hypertension. Am J Hypertens. 2025 Mar 17;38(4):248-256. doi: 10.1093/ajh/hpae152. PMID 39657776